CLINICAL TRIAL: NCT01090414
Title: An Extension Study to Investigate the Safety and Durability of Clinical Activity of Idelalisib in Subjects With Hematologic Malignancies
Brief Title: An Extension Study for Subjects Who Are Deriving Benefit With Idelalisib (GS-1101; CAL-101) Following Completion of a Prior Idelalisib Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-99
Record Dates: First submitted 2010-03-17; First posted 2010-03-22 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Lymphocytic Leukemia; Lymphoma, Non-Hodgkin
Keywords: Idelalisib; Chronic lymphocytic leukemia (CLL); Non-Hodgkin lymphoma (NHL); Phosphatidylinositol 3-kinase (PI3K)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idelalisib (Experimental): Participants will receive up to 350 mg of idelalisib twice daily until disease progression or unacceptable toxicity.
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib tablets or capsules administered orally
  Other Names: Zydelig®; GS-1101; CAL-101

SUMMARY:
This is a long-term safety extension study of idelalisib (GS-1101; CAL-101) in patients with hematologic malignancies who complete other idelalisib studies. It provides the opportunity for patients to continue treatment as long as the patient is deriving clinical benefit. Patients will be followed according to the standard of care as appropriate for their type of cancer. The dose of idelalisib will generally be the same as the dose that was administered at the end of the prior study, but may be titrated up to improve clinical response or down for toxicity. Patients will be withdrawn from the study if they develop progressive disease, unacceptable toxicity related to idelalisib, or if they no longer derive clinical benefit in the opinion of the investigator.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with hematologic malignancies completing a prior idelalisib study with a clinical benefit are eligible
* Women of childbearing potential must have a negative pregnancy test to be eligible
* Male patients, and female patients of childbearing potential, must agree to use method(s) of contraception specified in the protocol

Key Exclusion Criteria:

* Patients who are unwilling or unable to comply with the protocol are not eligible

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-03-22 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (18):
  - Clearview Cancer Institute, Huntsville, Alabama
  - UCLA, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Center for Cancer & Blood Disorders, PC, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Long Island Jewish medical Center, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer and Research Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Yakima Regional Cancer Care, Yakima, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Barrientos J, Coutre SE, et al. (2014). Long-Term Follow-Up of a Phase 1 Trial of Idelalisib (ZYDELIG®) in Combination with Bendamustine, Bendamustine/Rituximab, Fludarabine, Chlorambucil, or Chlorambucil/Rituximab in Patients with Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL) [Abstract 3343]. 56th American Society of Hematology (ASH) Annual Meeting and Exposition, San Francisco, California.
- [Result] Barrientos JC, Leonard JP, et al. (2013). Update on a Phase 1 Study of the Selective PI3Kδ Inhibitor, Idelalisib (GS-1101) in Combination with Rituximab and/or Bendamustine in Patients with Relapsed or Refractory CLL [Presentation]. American Society for Clinical Oncology (ASCO) Annual Meeting, Chicago, Illinois.
- [Result] Barrientos JC, Wagner-Johnston ND, et al. (2013). Chemo-Immunotherapy Combination of Idelalisib with Bendamustine/Rituximab or Chlorambucil/Rituximab in Patients with Relapsed/ Refractory CLL Demonstrates Efficacy and Tolerability [Poster 4176]. 55th ASH Annual Meeting and Exposition, New Orleans, Louisiana.
- [Result] Barrientos JC, Sharman J, et al. (2012). GS-1101 (CAL-101), A Selective Phosphatidylinositol 3-Kinase-Delta Inhibitor, in Combination With Ofatumumab for the Treatment of Relapsed/ Refractory CLL [Abstract 1062]. Haematologica: the Hematology Journal 17th Congress of the European Hematology Association 14-17 June 2012 Amsterdam; Netherlands 97 (Suppl 1): 433.
- [Result] Benson D, Kahl BS, et al. (2013). Final Results of a Phase 1 Study of Idelalisib, a Selective Inhibitor of PI3Kδ, in Patients with Relapsed or Refractory Indolent non-Hodgkin Lymphoma [Presentation]. ASCO Annual Meeting, Chicago, Illinois.
- [Result] Brown JR, Cheson BD, et al. (2015). Patterns of Lymphocytosis in Patients with CLL or Small Lymphocytic Lymphoma (SLL) Treated with Idelalisib. 57th ASH Annual Meeting and Exposition, Orlando, Florida.
- [Result] Brown JR, Byrd JC, Coutre SE, Benson DM, Flinn IW, Wagner-Johnston ND, Spurgeon SE, Kahl BS, Bello C, Webb HK, Johnson DM, Peterman S, Li D, Jahn TM, Lannutti BJ, Ulrich RG, Yu AS, Miller LL, Furman RR. Idelalisib, an inhibitor of phosphatidylinositol 3-kinase p110delta, for relapsed/refractory chronic lymphocytic leukemia. Blood. 2014 May 29;123(22):3390-7. doi: 10.1182/blood-2013-11-535047. Epub 2014 Mar 10. PMID 24615777
- [Result] Brown JR, Furman RR, et al. (2013). Final Results of a Phase 1 Study of Idelalisib (GS-1101) a Selective Inhibitor of Phosphatidylinositol 3-Kinase p110 Delta (PI3Kδ) in Patients with Relapsed or Refractory CLL [Presentation]. ASCO Annual Meeting, Chicago, Illinois.
- [Result] Coutre SE, Flinn IW, de Vos S, Barrientos JC, Schreeder MT, Wagner-Johnson ND, Sharman JP, Boyd TE, Fowler N, Dreiling L, Kim Y, Mitra S, Rai K, Leonard JP, Furman RR. Idelalisib in Combination With Rituximab or Bendamustine or Both in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia. Hemasphere. 2018 Apr 25;2(3):e39. doi: 10.1097/HS9.0000000000000039. eCollection 2018 Jun. PMID 31723767
- [Result] Coutre S, Barrientos C, et al. (2015). Safety of Idelalisib in B-cell Malignancies: Integrated Analysis of Eight Clinical Trials. ASCO Annual Meeting, Chicago, Illinois.
- [Result] Coutre S, Leonard J, et al. (2015). Idelalisib Monotherapy Results in Durable Responses in Patients with Relapsed or Refractory Waldenstrom's Macroglobulinemia. ASCO Annual Meeting, Chicago, Illinois.
- [Result] DeVos S, Wagner-Johnston ND, et al. (2014). Durable Responses Following Treatment with the PI3K-Delta Inhibitor Idelalisib in Combination with Rituximab, Bendamustine, or Both, in Recurrent Indolent non-Hodgkin Lymphoma: Phase I/II Results [Abstract 3063]. 56th ASH Annual Meeting and Exposition, San Francisco, California.
- [Result] DeVos S, Furman RR, et al. (2013). Idelalisib, a Selective Inhibitor of PI3Kδ, in Combination with Bendamustine, Fludarabine, or Chlorambucil in Patients with Relapsed or Refractory (R/R) CLL [Poster 2878]. 55th ASH Annual Meeting and Exposition, New Orleans, Louisiana.
- [Result] Flinn IW, Kahl BS, Leonard JP, Furman RR, Brown JR, Byrd JC, Wagner-Johnston ND, Coutre SE, Benson DM, Peterman S, Cho Y, Webb HK, Johnson DM, Yu AS, Ulrich RG, Godfrey WR, Miller LL, Spurgeon SE. Idelalisib, a selective inhibitor of phosphatidylinositol 3-kinase-delta, as therapy for previously treated indolent non-Hodgkin lymphoma. Blood. 2014 May 29;123(22):3406-13. doi: 10.1182/blood-2013-11-538546. Epub 2014 Mar 10. PMID 24615776
- [Result] Furman R, DeVos S, et al. (2014). Long-Term Follow-Up of a Phase 1 Study of Idelalisib (ZYDELIG®) in Combination with Anti-CD20 Antibodies (Rituximab or Ofatumumab) in Patients with Relapsed or Refractory CLL. 56th ASH Annual Meeting and Exposition, San Francisco, California.
- [Result] Furman R, Sharman J, et al. (2013). A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Idelalisib and Rituximab for Previously Treated Patients with CLL [Abstract LBA-6]. 55th ASH Annual Meeting and Exposition, New Orleans, Louisiana.
- [Result] Ghia P, Cheson BD, et al. (2016). Patterns of Idelalisib Treatment-Emergent Lymphocytosis in Patients with CLL or SLL [poster]. EHA 21st Congress, Copenhagen, Denmark.
- [Result] Ghia P, Coutre S, et al. (2016). Management of Transaminase Elevations Associated with Idelalisib [poster]. European Hematology Association (EHA) 21st Congress, Copenhagen, Denmark.
- [Result] Gopal AK, Davies AJ, et al. (2015). Idelalisib Monotherapy and Durable Responses in Patients with Relapsed or Refractory SLL. 57th ASH Annual Meeting and Exposition, Orlando, Florida.
- [Result] Kahl BS, Spurgeon SE, Furman RR, Flinn IW, Coutre SE, Brown JR, Benson DM, Byrd JC, Peterman S, Cho Y, Yu A, Godfrey WR, Wagner-Johnston ND. A phase 1 study of the PI3Kdelta inhibitor idelalisib in patients with relapsed/refractory mantle cell lymphoma (MCL). Blood. 2014 May 29;123(22):3398-405. doi: 10.1182/blood-2013-11-537555. Epub 2014 Mar 10. PMID 24615778
- [Result] Leonard JP, Wagner-Johnston ND, et al. (2013). Combinations of the PI3Kδ Inhibitor Idelalisib (GS-1101) with Rituximab and/or Bendamustine are Tolerable and Highly Active in Patients with Previously Treated, Indolent non-Hodgkin Lymphoma: Updated Results from a Phase I Study [Presentation]. ASCO Annual Meeting, Chicago, Illinois.
- [Result] Martin P, Armas A, et al. (2015). Idelalisib Monotherapy and Durable Responses in Patients with Relapsed or Refractory Marginal Zone Lymphoma (MZL). 57th ASH Annual Meeting and Exposition, Orlando, Florida.
- [Result] O'Brien SM, Lamanna N, Kipps TJ, Flinn I, Zelenetz AD, Burger JA, Keating M, Mitra S, Holes L, Yu AS, Johnson DM, Miller LL, Kim Y, Dansey RD, Dubowy RL, Coutre SE. A phase 2 study of idelalisib plus rituximab in treatment-naive older patients with chronic lymphocytic leukemia. Blood. 2015 Dec 17;126(25):2686-94. doi: 10.1182/blood-2015-03-630947. Epub 2015 Oct 15. PMID 26472751
- [Result] O'Brien SM, Lamanna N, et al. (2014). Update on a Phase 2 Study of Idelalisib in Combination with Rituximab in Treatment-Naive Patients ≥ 65 Years with CLL or SLL [Poster 1994]. 56th ASH Annual Meeting and Exposition, San Francisco, California.
- [Result] O'Brien SM, Lamanna N, et al. (2013). A Phase 2 Study of the Selective Phosphatidylinositol 3-Kinase Delta (PI3Kδ) Inhibitor Idelalisib (GS-1101) in Combination with Rituximab in Treatment-Naive Patients ≥ 65 Years with CLL or SLL [Presentation]. ASCO Annual Meeting, Chicago, Illinois.
- [Result] Spurgeon SE, Wagner-Johnston ND, et al. (2013). Final Results of a Phase 1 Study of Idelalisib, a Selective Inhibitor of Phosphatidylinositol 3-Kinase P110δ (PI3Kδ) in Patients with Relapsed or Refractory Mantle Cell Lymphoma [Presentation]. ASCO Annual Meeting, Chicago, Illinois.
- [Result] Wagner-Johnston ND, DeVos S, et al. (2013). Preliminary Results of PI3Kδ Inhibitor Idelalisib (GS-1101) Treatment in Combination with Everolimus, Bortezomib, or Bendamustine/Rituximab in Patients with Previously Treated Mantle Cell Lymphoma [Presentation]. ASCO Annual Meeting, Chicago, Illinois.
- [Result] Wierda W, Coutre S, et al. (2016). Management of Transaminase Elevations in Patients Receiving Idelalisib. ASCO Annual Meeting, Chicago, Illinois.
- [Derived] de Vos S, Wagner-Johnston ND, Coutre SE, Flinn IW, Schreeder MT, Fowler NH, Sharman JP, Boccia RV, Barrientos JC, Rai KR, Boyd TE, Furman RR, Kim Y, Godfrey WR, Leonard JP. Combinations of idelalisib with rituximab and/or bendamustine in patients with recurrent indolent non-Hodgkin lymphoma. Blood Adv. 2016 Nov 30;1(2):122-131. doi: 10.1182/bloodadvances.2016000976. eCollection 2016 Dec 13. PMID 29296805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 22 March 2010. The last study visit occurred on 18 June 2018.
Pre-assignment Details: Participants must have been enrolled in a previous Gilead-sponsored study.
Groups:
- 101-02: Participants with chronic lymphocytic leukemia (CLL), indolent non-Hodgkin lymphoma (iNHL), mantle cell lymphoma (MCL), diffuse large B-cell lymphoma (DLBCL), acute myeloid leukemia (AML), or multiple myeloma (MM) received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-07: Participants with CLL, iNHL, or MCL received idelalisib 100 mg or 150 mg tablets twice daily with or without rituximab, bendamustine, ofatumumab, fludarabine, everolimus, bortezomib, chlorambucil, and/or lenalidomide during parent study 101-07 (NCT01088048, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-08: Participants with CLL or iNHL (specifically, small lymphocytic lymphoma (SLL)) received idelalisib 150 mg tablets twice daily with rituximab during parent study 101-08 (NCT01203930) and may have entered long-term safety extension study 101-99 to receive the same treatment. Note: Only participants from Cohort 1 were eligible to enter this Study 101-99, so Cohort 2 participants are not presented at all in this record.
- 101-10: Participants with iNHL received idelalisib 150 mg tablets twice daily during parent study 101-10 (NCT01306643) and may have entered long-term safety extension study 101-99 to receive the same treatment.
Period: Parent Studies
Arm/Group | 101-02 | 101-07 | 101-08 | 101-10
Started | 191 | 241 | 64 | 18
Completed (Study completion was defined as participants who completed through Week 48 of parent study.) | 50 | 114 | 43 | 5
Not Completed | 141 | 127 | 21 | 13
Period: Study 101-99
Arm/Group | 101-02 | 101-07 | 101-08 | 101-10
Started | 48 (50 participants completed the parent study, but only 48 participants enrolled into Study 101-99.) | 108 (114 participants completed the parent study, but only 108 participants enrolled into Study 101-99.) | 41 (43 participants completed the parent study, but only 41 participants enrolled into Study 101-99.) | 5
Completed | 0 | 0 | 0 | 0
Not Completed | 48 | 108 | 41 | 5
Not completed — Progressive Disease | 28 | 48 | 10 | 4
Not completed — Adverse Event | 10 | 28 | 18 | 0
Not completed — Investigator Request | 1 | 11 | 4 | 0
Not completed — Death | 3 | 8 | 1 | 0
Not completed — Sponsor Discontinued Study | 0 | 7 | 5 | 0
Not completed — Other (Unknown Reasons) | 3 | 3 | 0 | 0
Not completed — Withdrew Consent | 0 | 2 | 3 | 1
Not completed — Participant Request | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data presented includes baseline characteristic data for all participants who received any dose of idelalisib in the parent studies, excluding Cohort 2 participants from Study 101-08 who were not eligible to enroll into Study 101-99.
Groups:
- 101-02: Participants with CLL, iNHL, MCL, DLBCL, AML, or MM received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-08: Participants with CLL or iNHL (specifically, small lymphocytic lymphoma (SLL)) received idelalisib 150 mg tablets twice daily with rituximab during parent study 101-08 (NCT01203930) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- Total: Total of all reporting groups
Arm/Group | 101-02 | 101-07 | 101-08 | 101-10 | Total
Number analyzed (Participants) | 191 | 241 | 64 | 18 | 514
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 86 | 116 | 0 | 13 | 215
  ≥ 65 years | 105 | 125 | 64 | 5 | 299
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 76 | 24 | 8 | 160
  Male | 139 | 165 | 40 | 10 | 354
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 0 | 1 | 7
  Not Hispanic or Latino | 167 | 234 | 64 | 17 | 482
  Unknown or Not Reported | 22 | 3 | 0 | 0 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 160 | 209 | 61 | 12 | 442
  Race: Black or African American | 6 | 9 | 1 | 5 | 21
  Race: Asian | 1 | 11 | 1 | 1 | 14
  Race: Other | 2 | 1 | 1 | 0 | 4
  Race: Not Reported | 22 | 11 | 0 | 0 | 33
Diagnosis Status [Count of Participants; unit: Participants] — Diagnosis status of iNHL included the following types: follicular lymphoma (FL), small lymphocytic lymphoma (SLL), lymphoplasmacytic lymphoma/Waldenstrom's Macroglobulinemia (LPL/WM), and marginal zone lymphoma (MZL).
  Participants
    Chronic lymphocytic leukemia (CLL) | 54 | 115 | 59 | 0 | 228
    Indolent non-Hodgkin lymphoma (iNHL) | 64 | 86 | 5 | 17 | 172
    Mantle cell lymphoma (MCL) | 40 | 40 | 0 | 0 | 80
    Diffuse large B-cell lymphoma (DLBCL) | 9 | 0 | 0 | 0 | 9
    Acute myeloid leukemia (AML) | 12 | 0 | 0 | 0 | 12
    Multiple myeloma (MM) | 12 | 0 | 0 | 0 | 12
    Missing | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) was defined as the percentage of participants who achieve complete response (CR), partial response (PR), or minor response (MR; for lymphoplasmacytic lymphoma/Waldenström's macroglobulinemia (LPL/WM) only).
Time Frame: Parent study baseline to end of study 101-99 (maximum: up to 91.2 months)
Population: Data presented includes available data from both the parent studies and this Study 101-99. It was prespecified that data for Study 101-08 be combined for CLL and SLL participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 101-02 (AML): Participants with AML received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-02 (CLL): Participants with CLL received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-02 (DLBCL): Participants with DLBCL received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-02 (iNHL): Participants with iNHL received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-02 (MCL): Participants with MCL received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-02 (MM): Participants with MM received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-07 (CLL): Participants with CLL received idelalisib 100 mg or 150 mg tablets twice daily with or without rituximab, bendamustine, ofatumumab, fludarabine, chlorambucil, and/or lenalidomide during parent study 101-07 (NCT01088048, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-07 (iNHL): Participants with iNHL received idelalisib 100 mg or 150 mg tablets twice daily with or without rituximab, bendamustine, and/or lenalidomide during parent study 101-07 (NCT01088048, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-07 (MCL): Participants with MCL received idelalisib 100 mg or 150 mg tablets twice daily with or without rituximab, bendamustine, everolimus, bortezomib, and/or lenalidomide during parent study 101-07 (NCT01088048, results reported within this record) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-08 (CLL or SLL): Participants with CLL or SLL received idelalisib 150 mg tablets twice daily with rituximab during parent study 101-08 (NCT01203930) and may have entered long-term safety extension study 101-99 to receive the same treatment.
- 101-10 (iNHL): Participants with iNHL received idelalisib 150 mg tablets twice daily during parent study 101-10 (NCT01306643) and may have entered long-term safety extension study 101-99 to receive the same treatment.
Arm/Group | 101-02 (AML) | 101-02 (CLL) | 101-02 (DLBCL) | 101-02 (iNHL) | 101-02 (MCL) | 101-02 (MM) | 101-07 (CLL) | 101-07 (iNHL) | 101-07 (MCL) | 101-08 (CLL or SLL) | 101-10 (iNHL)
Number analyzed (Participants) | 12 | 54 | 9 | 64 | 40 | 12 | 115 | 86 | 40 | 64 | 18
percentage of participants | 0 [0 to 0] | 57.4 [43.2 to 70.8] | 11.1 [0.3 to 48.2] | 48.4 [35.8 to 61.3] | 40.0 [24.9 to 56.7] | 0 [0 to 0] | 81.7 [73.5 to 88.3] | 82.6 [72.9 to 89.9] | 57.5 [40.9 to 73.0] | 96.9 [89.2 to 99.6] | 44.4 [21.5 to 69.2]

2. Primary Outcome: Percentage of Participants Who Experienced Any Treatment-Emergent Adverse Events
Time Frame: Parent study baseline to end of study 101-99 (maximum: up to 91.2 months) plus 30 days
Population: Data presented includes data from both the parent studies and this Study 101-99. For this safety endpoint, data was prespecified to be combined.
Measure: Number; unit: percentage of participants
Groups:
- 101-02: Participants with CLL or iNHL received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and entered long-term safety extension study 101-99 to receive the same treatment.
- 101-07: Participants with CLL, iNHL, or MCL received idelalisib 100 mg or 150 mg tablets twice daily with or without rituximab, bendamustine, ofatumumab, fludarabine, everolimus, bortezomib, chlorambucil, and/or lenalidomide during parent study 101-07 (NCT01088048, results reported within this record) and entered long-term safety extension study 101-99 to receive the same treatment.
- 101-08: Participants with CLL or SLL received idelalisib 150 mg tablets twice daily with rituximab during parent study 101-08 (NCT01203930) and entered long-term safety extension study 101-99 to receive the same treatment.
- 101-10: Participants with iNHL received idelalisib 150 mg tablets twice daily during parent study 101-10 (NCT01306643) and entered long-term safety extension study 101-99 to receive the same treatment.
Arm/Group | 101-02 | 101-07 | 101-08 | 101-10
Number analyzed (Participants) | 191 | 241 | 64 | 18
percentage of participants | 98.4 | 98.8 | 100.0 | 94.4

3. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the interval from the first documentation of CR, PR, or MR (for LPL/WM) to the earlier of the first documentation of disease progression or death from any cause. DOR was analyzed using Kaplan-Meier (KM) estimates.
Time Frame: Parent study baseline to end of study 101-99 (maximum: up to 91.2 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 101-02 (AML) | 101-02 (CLL) | 101-02 (DLBCL) | 101-02 (iNHL) | 101-02 (MCL) | 101-02 (MM) | 101-07 (CLL) | 101-07 (iNHL) | 101-07 (MCL) | 101-08 (CLL or SLL) | 101-10 (iNHL)
Number analyzed (Participants) | 12 | 54 | 9 | 64 | 40 | 12 | 115 | 86 | 40 | 64 | 18
Months | NA [NA to NA] — NA = No participants achieved complete or partial response. | 21.2 [8.1 to 30.4] | NA [NA to NA] — NA = not reached; Too few events to estimate the median and the lower and upper limits of the confidence interval. | 18.4 [10.9 to 32.4] | 2.7 [1 to 8.1] | NA [NA to NA] — NA = No participants achieved complete or partial response. | 26.6 [18.5 to 44.1] | 42.9 [20.5 to 83.3] | 9.3 [5.6 to 37.5] | 63.8 [54.0 to NA] — NA = Not reached; Too few events to estimate the upper limit of the confidence interval. | 14.4 [6.6 to 46.3]

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the interval from start of idelalisib treatment in the parent study to the earlier of the first documentation of disease progression or death from any cause. PFS was analyzed using KM estimates.
Time Frame: Parent study baseline to end of study 101-99 (maximum: up to 91.2 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 101-02 (AML) | 101-02 (CLL) | 101-02 (DLBCL) | 101-02 (iNHL) | 101-02 (MCL) | 101-02 (MM) | 101-07 (CLL) | 101-07 (iNHL) | 101-07 (MCL) | 101-08 (CLL or SLL) | 101-10 (iNHL)
Number analyzed (Participants) | 12 | 54 | 9 | 64 | 40 | 12 | 115 | 86 | 40 | 64 | 18
Months | 0.9 [0.4 to 1] | 15.8 [5.6 to 39.6] | 1.5 [0.3 to 4.1] | 7.6 [3.7 to 17.7] | 3.7 [2.7 to 8.2] | 1 [0.9 to 1.8] | 26.1 [19.0 to 36.8] | 32.8 [22.0 to 81.3] | 11.1 [3.4 to 12.9] | 65.6 [55.8 to NA] — NA = Not reached; Too few events to estimate the upper limit of the confidence interval. | 10.2 [2.8 to 19.1]

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the interval from the start of study treatment in the parent study to death from any cause. OS was analyzed using KM estimates.
Time Frame: Parent study baseline to end of study 101-99 (maximum: up to 91.2 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 101-02 (AML) | 101-02 (CLL) | 101-02 (DLBCL) | 101-02 (iNHL) | 101-02 (MCL) | 101-02 (MM) | 101-07 (CLL) | 101-07 (iNHL) | 101-07 (MCL) | 101-08 (CLL or SLL) | 101-10 (iNHL)
Number analyzed (Participants) | 12 | 54 | 9 | 64 | 40 | 12 | 115 | 86 | 40 | 64 | 18
Months | NA [NA to NA] — NA = not reached; Too few events to estimate the median and the lower and upper limits of the confidence interval. | NA [39.7 to NA] — NA = not reached; Too few events to estimate the median and upper limit of the confidence interval. | NA [NA to NA] — NA = not reached; Too few events to estimate the median and the lower and upper limits of the confidence interval. | NA [NA to NA] — NA = not reached; Too few events to estimate the median and the lower and upper limits of the confidence interval. | NA [NA to NA] — NA = not reached; Too few events to estimate the median and the lower and upper limits of the confidence interval. | 5.2 [1.2 to 5.2] | NA [50.2 to NA] — NA = not reached; Too few events to estimate the median and upper limit of the confidence interval. | NA [NA to NA] — NA = not reached; Too few events to estimate the median and the lower and upper limits of the confidence interval. | NA [NA to NA] — NA = not reached; Too few events to estimate the median and the lower and upper limits of the confidence interval. | NA [66.3 to NA] — NA = not reached; Too few events to estimate the median and upper limit of the confidence interval. | NA [10.3 to NA] — NA = not reached; Too few events to estimate the median and upper limit of the confidence interval.

6. Secondary Outcome: Time to Response
Description: Time to response (TTR) was defined as the interval from start of study treatment to the first documentation of CR, PR, or MR (for LPL/WM). Analysis only includes participants who achieved complete or partial response (or minor response for LPL/WM participants). No participants in the 101-02 (AML and MM) groups achieved a complete or partial response.
Time Frame: Parent study baseline to end of study 101-99 (maximum: up to 91.2 months)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Groups:
- 101-10 (iNHL): Participants iNHL received idelalisib 150 mg tablets twice daily during parent study 101-10 (NCT01306643) and may have entered long-term safety extension study 101-99 to receive the same treatment.
Arm/Group | 101-02 (AML) | 101-02 (CLL) | 101-02 (DLBCL) | 101-02 (iNHL) | 101-02 (MCL) | 101-02 (MM) | 101-07 (CLL) | 101-07 (iNHL) | 101-07 (MCL) | 101-08 (CLL or SLL) | 101-10 (iNHL)
Number analyzed (Participants) | 0 | 31 | 1 | 31 | 16 | 0 | 94 | 71 | 23 | 62 | 8
Months |  | 1.9 [1.0 to 7.5] | 4.0 [4.0 to 4.0] | 1.3 [1.0 to 3.7] | 1.1 [1.0 to 1.9] |  | 1.9 [1.9 to 1.9] | 1.9 [1.9 to 3.0] | 1.9 [1.9 to 2.0] | 1.9 [1.9 to 1.9] | 2.7 [2.6 to 3.1]

ADVERSE EVENTS:
Time Frame: First dose date in parent study to end of study 101-99 (maximum: up to 91.2 months) plus 30 days
Description: Adverse events presented occurred during either the parent studies or Study 101-99. Because Study 101-99 was a long-term extension study, the adverse event data was prespecified to be combined and reported based on the participation in the parent studies.
Groups:
- 101-02: Participants with CLL, iNHL, MCL, DLBCL, AML, or MM received idelalisib 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, or 350 mg capsules twice daily during parent study 101-02 (NCT00710528, results reported within this record) and may have entered the long-term safety extension study 101-99 to receive the same treatment.
- 101-08: Participants with CLL or SLL received idelalisib 150 mg tablets twice daily with rituximab during parent study 101-08 (NCT01203930) and may have entered long-term safety extension study 101-99 to receive the same treatment.
Arm/Group | 101-02 | 101-07 | 101-08 | 101-10
All-Cause Mortality (participants affected / at risk) | 25/191 | 36/241 | 7/45 | 2/6
Serious Adverse Events (participants affected / at risk) | 100/191 | 165/241 | 45/64 | 6/18
Other Adverse Events (participants affected / at risk) | 183/191 | 236/241 | 63/64 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 101-02 (N=191) | 101-07 (N=241) | 101-08 (N=64) | 101-10 (N=18)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 1 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Autoimmune neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Coombs positive haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 12 | 23 | 3 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 6 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 4 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Endocrine disorder (Endocrine disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Colitis (Gastrointestinal disorders) | 8 | 14 | 13 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 14 | 13 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 6 | 31 | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abdominal wall infection (Infections and infestations) | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 2 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 2 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 4 | 2 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Cerebral aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 1 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1 | 0
Corynebacterium bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 1 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 2 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 2 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 4 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Histoplasmosis (Infections and infestations) | 0 | 1 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 0 | 2 | 0 | 0
Hydrocele male infected (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 2 | 1 | 0
Listeria sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Listeriosis (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis enterococcal (Infections and infestations) | 1 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 2 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 8 | 1 | 0
Pneumonia (Infections and infestations) | 30 | 40 | 12 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 3 | 3 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 3 | 2 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 4 | 14 | 1 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 2 | 0 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 3 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Vulvovaginitis (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 4 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 1 | 0
Liver function test increased (Investigations) | 2 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 3 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 4 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 9 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 0 | 0 | 2
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 4 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Vasculitis necrotising (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 101-02 (N=191) | 101-07 (N=241) | 101-08 (N=64) | 101-10 (N=18)
Anaemia (Blood and lymphatic system disorders) | 31 | 48 | 7 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 21 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 31 | 102 | 5 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 48 | 3 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 8 | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 6 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 7 | 1 | 2
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 1
Chalazion (Eye disorders) | 0 | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 5 | 7 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 5 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 31 | 8 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7 | 5 | 0
Colitis (Gastrointestinal disorders) | 3 | 8 | 3 | 1
Constipation (Gastrointestinal disorders) | 23 | 49 | 11 | 3
Diarrhoea (Gastrointestinal disorders) | 58 | 106 | 36 | 8
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 15 | 3 | 0
Flatulence (Gastrointestinal disorders) | 8 | 9 | 4 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 11 | 4 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Lip discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 44 | 81 | 24 | 7
Oral pain (Gastrointestinal disorders) | 2 | 3 | 1 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 10 | 18 | 8 | 0
Vomiting (Gastrointestinal disorders) | 23 | 33 | 14 | 5
Asthenia (General disorders) | 16 | 21 | 7 | 2
Chest discomfort (General disorders) | 1 | 5 | 4 | 0
Chest pain (General disorders) | 1 | 9 | 0 | 1
Chills (General disorders) | 31 | 40 | 23 | 2
Fatigue (General disorders) | 63 | 85 | 21 | 8
Influenza like illness (General disorders) | 0 | 2 | 9 | 2
Malaise (General disorders) | 1 | 4 | 6 | 2
Mucosal inflammation (General disorders) | 7 | 15 | 0 | 0
Oedema (General disorders) | 3 | 8 | 4 | 0
Oedema peripheral (General disorders) | 18 | 29 | 7 | 0
Pain (General disorders) | 6 | 24 | 1 | 2
Pyrexia (General disorders) | 49 | 92 | 26 | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 4 | 0 | 1
Candida infection (Infections and infestations) | 5 | 5 | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 4 | 1 | 1
Herpes zoster (Infections and infestations) | 4 | 13 | 2 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 5 | 11 | 3 | 2
Pneumonia (Infections and infestations) | 6 | 18 | 7 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 10 | 22 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 32 | 38 | 8 | 4
Urinary tract infection (Infections and infestations) | 10 | 15 | 9 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 2 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 5 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 14 | 7 | 0
Alanine aminotransferase increased (Investigations) | 33 | 52 | 18 | 8
Aspartate aminotransferase increased (Investigations) | 35 | 47 | 18 | 8
Blood alkaline phosphatase increased (Investigations) | 12 | 13 | 2 | 0
Blood bilirubin increased (Investigations) | 2 | 6 | 1 | 2
Blood creatinine increased (Investigations) | 11 | 9 | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 4 | 14 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 1
Liver function test increased (Investigations) | 6 | 5 | 6 | 0
Neutrophil count decreased (Investigations) | 8 | 9 | 5 | 1
Transaminases increased (Investigations) | 6 | 5 | 9 | 4
Weight decreased (Investigations) | 10 | 21 | 7 | 2
Decreased appetite (Metabolism and nutrition disorders) | 22 | 41 | 9 | 3
Dehydration (Metabolism and nutrition disorders) | 11 | 10 | 6 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 12 | 4 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 10 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 12 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 35 | 6 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 11 | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 16 | 7 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 9 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 16 | 10 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 24 | 9 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 5 | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 10 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 13 | 6 | 3
Dizziness (Nervous system disorders) | 15 | 32 | 7 | 0
Dysgeusia (Nervous system disorders) | 6 | 24 | 4 | 3
Headache (Nervous system disorders) | 22 | 31 | 15 | 4
Hypersomnia (Nervous system disorders) | 0 | 1 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 2 | 0 | 2
Mental impairment (Nervous system disorders) | 0 | 2 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 9 | 2 | 1
Agitation (Psychiatric disorders) | 0 | 2 | 1 | 2
Anxiety (Psychiatric disorders) | 5 | 16 | 4 | 0
Confusional state (Psychiatric disorders) | 4 | 3 | 1 | 1
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 17 | 36 | 13 | 5
Acute kidney injury (Renal and urinary disorders) | 4 | 7 | 4 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 3 | 7 | 2 | 1
Nocturia (Renal and urinary disorders) | 2 | 4 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 5 | 3 | 2 | 1
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 81 | 21 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 42 | 14 | 2
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 12 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 18 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 20 | 4 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 1 | 4 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 23 | 23 | 10 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 29 | 11 | 3
Rash (Skin and subcutaneous tissue disorders) | 39 | 65 | 24 | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 4 | 10 | 4 | 0
Hot flush (Vascular disorders) | 1 | 2 | 2 | 1
Hypertension (Vascular disorders) | 6 | 11 | 4 | 0
Hypotension (Vascular disorders) | 8 | 7 | 7 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (8):
  • Study Protocol: Original (2010-01-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT01090414/Prot_000.pdf
  • Study Protocol: Amendment 1 (2010-04-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT01090414/Prot_001.pdf
  • Study Protocol: Amendment 2 (2013-10-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT01090414/Prot_002.pdf
  • Study Protocol: Amendment 3 (2014-11-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT01090414/Prot_003.pdf
  • Study Protocol: Amendment 4 (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT01090414/Prot_004.pdf
  • Study Protocol: Amendment 5 (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT01090414/Prot_005.pdf
  • Study Protocol: Amendment 6 (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT01090414/Prot_006.pdf
  • Statistical Analysis Plan (2013-04-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT01090414/SAP_007.pdf